CLINICAL TRIAL: NCT03934905
Title: Phase II Trial of Effects of the Nutritional Supplement Sulforaphane on Doxorubicin-Associated Cardiac Dysfunction (CRI18-026)
Brief Title: Protective Effects of the Nutritional Supplement Sulforaphane on Doxorubicin-Associated Cardiac Dysfunction
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: L19-065
Record Dates: First submitted 2019-03-29; First posted 2019-05-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Anthracycline Related Cardiotoxicity in Breast Cancer
Keywords: doxorubicin; sulforaphane; cardiotoxicity; nrf2; heart
MeSH Terms: conditions — Cardiotoxicity | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: We plan to include 70 DOX-naïve women with breast cancer undergoing neoadjuvant chemotherapy, with no prior cardiac disease and who will receive DOX without Her-2 receptor antagonists as part of their clinical care. Potential subjects will be recruited in a randomized, controlled; double blinded pilot study comparing SFN to placebo. Study will be conducted at the TTUHSC and UMC. The trial is approved by the institutional IRB and will be registered at clinicaltrials.gov. UMC cancer center pharmacist Ajoke A. Tijani, RPh. will receive placebo and test compound from supplier and will dispense them to test subjects. Randomization will be done with assignment of a subject ID to the study subject. The list of subject IDs will be subsequently assigned to either study drug or placebo using a randomizer software.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sulforaphane (Active Comparator): Processed SFN-rich extract will be purchased in form of caplets from Nutramax Laboratories, Inc. 2208 Lakeside Blvd Edgewood, MD 21040. Caplets containing SFN-rich broccoli sprout extracts from Nutramax Labs will be dispensed to participants in sealed bottles with instructions to keep them in a household freezer. Size of the caplet will be about 2 cm in length. Dosing will be based on weight and will be dosed daily for 12 weeks.
  Interventions: Drug: sulforaphane
- Placebo (Placebo Comparator): Placebo caplets will comprise of microcrystalline cellulose from Nutramax Labs and will be dispensed to participants in sealed bottles with instructions to keep them in a household freezer. Placebo pills will be identical in appearance to the sulforaphane pills and will be dosed in a similar manner (identical number of pills based on weight, daily dosing and for 12 weeks)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: sulforaphane — The participants will be dosed, based on weight, in a double-blind fashion with identical appearing placebo or sulforaphane caplets in a daily dose for 12 weeks of: two caplets for individuals <100 lb., four caplets for individuals 100-200 lb. and eight caplets for individuals >200 lb. Avmacol or placebo will be prescribed by Dr. Awasthi and will be dispensed by local pharmacy or study coordinators at TTUHSC/UMC Lubbock. We will be doing pill counts to make sure that volunteers have used as directed. We will measure the Sulforaphane level in plasma by well-established method.
  Arms: sulforaphane
Drug: Placebo Oral Tablet — The participants will be dosed, based on weight, in a double-blind fashion with identical appearing placebo or sulforaphane caplets in a daily dose for 12 weeks of: two caplets for individuals <100 lb., four caplets for individuals 100-200 lb. and eight caplets for individuals >200 lb. Avmacol or placebo will be prescribed by Dr. Awasthi and will be dispensed by local pharmacy or study coordinators at TTUHSC/UMC Lubbock. We will be doing pill counts to make sure that volunteers have used as directed. We will measure the Sulforaphane level in plasma by well-established method.
  Arms: Placebo

SUMMARY:
Cardiomyopathy is a major complication of doxorubicin (DOX) chemotherapy, and 10-21% of breast cancer patients receiving DOX experience compromised cardiac function. Recent advancements have increased cancer survivorship but it remains clinically challenging to mitigate the cardiotoxic side effects. Although there are several strategies used to reduce the occurrence and severity of DOX-induced cardiotoxicity, they are not particularly effective. Hence, there is an urgent need to develop new strategies that prevent the cardiotoxic effects of DOX but maintain its potency as a cancer therapy. Because the cellular events responsible for the antitumor activity of DOX and DOX-induced cardiotoxicity are distinctly different, it may be possible to develop therapies that selectively mitigate DOX-induced cardiotoxicity. Thus, the investigators propose to test an adjuvant therapy that combines the phytochemical sulforaphane (SFN) with DOX to attenuate DOX-induced cardiomyopathy. SFN activates the transcription factor Nrf2 and induces defense mechanisms in normal cells. Furthermore, SFN inhibits carcinogenesis and metastases and enhances cancer cell sensitivity to DOX, seemingly through Nrf2-independent mechanisms. SFN has also been tested in several clinical trials, although never together with DOX. Our early animal studies suggest that by activating Nrf2, SFN selectively protects the mouse and rat from DOX cardiotoxicity, enhances survival and enhances the effects of DOX on cancer growth in a rat breast cancer model. The investigators suspect that SFN affects DOX metabolism in cancer cells to enhance tumor regression, or it may synergistically activate other key antitumor mechanisms. Hence, SFN may improve the clinical outcome of cancer therapy by (1) attenuating DOX cardiotoxicity and (2) enhancing the effects of cancer treatment on the tumor. Our hypothesis is that SFN protects the heart from DOX-mediated cardiac injury without altering the antitumor efficacy of DOX. In Aim 1, the investigators will conduct an early-phase clinical trial to determine if SFN is safe to administer to breast cancer patients undergoing DOX chemotherapy. In Aim 2, the investigators will determine if SFN decreases DOX-induced inflammatory responses and enhances Nrf2- and SIRT1-target gene expression in breast cancer patients. Notably, transcript and protein signatures in peripheral blood mononuclear cells (PBMCs) can predict cardiac function in patients undergoing DOX chemotherapy for breast cancer. The investigators will also determine if SFN/DOX treatment activates Nrf2- and SIRT1-dependent gene expression, alters the levels of biomarkers for presymptomatic DOX-cardiotoxicity and mitigates the generation of cardiotoxic metabolites in PBMCs and plasma. These studies will facilitate the development of SFN co-treatment as a strategy to enhance the efficacy and safety of DOX cancer therapy.

DETAILED DESCRIPTION:
Determine whether nutritional supplement sulforaphane (SFN) is safe to administer to breast cancer patients undergoing doxorubicin (DOX) chemotherapy. The investigators have identified biomarkers for presymptomatic detection of DOX cardiotoxicity in breast cancer patients and reported that SFN alleviates DOX-induced cardiac toxicity while maintaining its anti-tumor activity in an animal model of breast cancer. SFN is in various stages of preclinical and clinical trials against different types of cancer but its safety and effects on identified markers have never been tested in patients treated with DOX. Sulforaphane is a generally recognized as a safe (GRAS) compound and this compound is currently in 61 different clinical trials including, Cystic Fibrosis, COPD, Melanoma, Breast and prostate cancer etc. (https://clinicaltrials.gov/ct2/results?term=sulforaphane&pg=1). Avmacol Extra Strength, (Nutramax Laboratories Consumer Care, Inc. Edgewood, MD 21040) an over-the-counter dietary supplement containing broccoli seed and sprout extracts that is rich with sulforaphane, will be used in this study. This is an FDA regulated trial using an investigational drug under IND 141682. Dose considerations were made on the basis of the ongoing clinical trial "Effects of Avmacol Extra Strength® in the Oral Mucosa of Patients Following Curative Treatment for Tobacco-related Head and Neck Cancer" (https://clinicaltrials.gov/ct2/show/NCT03268993). Furthermore, Avmacol Extra Strength has never been tested as an adjuvant to try and protect the heart from DOXs harmful effects. . Therefore, the investigators are proposing to do an early-clinical trial to assess SFN safety in DOX-treated patients and possibly prevent DOX-cardiotoxicity in breast cancer patients.

Our hypothesis is that SFN protects the heart from DOX-mediated cardiac injury without affecting its antitumor efficacy. Here, the investigators will test SFN in combination with DOX-based chemotherapy for breast cancer; the investigators will assess its safety, cardio-protective properties, and anti-cancer efficacy. The investigators will also examine the effect of SFN on the expression of several biomarkers that indicate when a patient cannot tolerate DOX.1 To test our hypothesis, the investigators propose the following Specific Aims.

Aim 1: Demonstrate that co-administration of SFN protects the heart and is not associated with toxicity or reduced tumor response in breast cancer patients undergoing DOX chemotherapy.

The investigators propose a pilot clinical trial to assess the safety of SFN as a co-treatment with DOX chemotherapy. Strategy: Up to seventy breast cancer patients prescribed DOX chemotherapy will be consented then randomly assigned to receive either SFN or placebo during DOX chemotherapy. This sample size includes an additional 10 participants to allow for potential attrition. There will be a 50-50 chance of receiving SFN. The patients will be recruited from the Breast Cancer Clinic (Dr. Jones and Philipovskiy) in the Southwest Cancer Center at TTUHSC/UMC Lubbock. Cardiac function with echocardiography will be assessed and compared between arms for evidence of substantive decrease in DOX cardiotoxicity with SFN compared to placebo. Tumor size will also be compared (based on RECIST criteria) between treatment arms. The investigators will monitor treatment-emergent symptoms, hematological parameters of cancer therapy toxicity, and renal and hepatic function. Blood samples will be collected to assay markers of cardiotoxicity, including B-type natriuretic peptide and troponin.

Aim 2: Determine if SFN alters the levels of known biomarkers of DOX cardiotoxicity and affects the expression of SIRT1- and Nrf2-target genes.

The investigators will measure changes in transcript and protein biomarkers of pre-symptomatic DOX-cardiotoxicity in response to SFN, and will determine if SFN promotes SIRT1- and Nrf2-dependent gene expression. Because Nrf2 upregulates certain detoxifying enzymes, the investigators will measure the plasma levels of cardiotoxic metabolites, doxorubicinol (DOXol). Strategy: Blood will be collected before the start of DOX chemotherapy and after each treatment cycle to isolate peripheral blood mononuclear cells (PBMCs) and prepare plasma. In lieu of tissue biopsies, PBMCs will be used to examine SIRT1 and Nrf2 activity and target gene expression. Multiplex arrays will be used to measure plasma cytokine levels, and plasma DOX metabolites will be assessed with ultrahigh performance liquid chromatography-tandem mass spectrometry. These experiments will provide initial evidence to indicate that SFN activates SIRT1 and Nrf2 pathways in non-cancer tissue of breast cancer patients.

Impact: This will be the first clinical study to assess the safety of SFN as a co-treatment with DOX to mitigate cardiotoxicity in breast cancer patients. Positive findings will be used to justify a larger randomized controlled trial. Subjects will be randomized at a 1:1 ratio.

Study Design and Procedures Study Design. The investigators intend to include up to 70 DOX-naïve women diagnosed with breast cancer undergoing neoadjuvant chemotherapy with no prior cardiac disease and who will receive DOX without Her-2 receptor antagonists (to eliminate possibility of secondary side effects) as part of their clinical care. These potential subjects will be recruited in a randomized, controlled, double blinded pilot study comparing SFN to placebo. The study will be conducted at the Texas Tech University Health Sciences Center, and University Medical Center. The trial will be approved by our local IRB and registered at clinicaltrials.gov. UMC cancer center pharmacist Ajoke A. Tijani, RPh. (Tijani@umchealthsystem.com) will receive placebo and test compound from supplier and will dispense them to test subjects.

Randomization will be achieved with assignment of a subject ID to the study subject. The list of subject IDs will be subsequently assigned either study drug or placebo using a randomizer software such as (www.randomizer.org). The pharmacist dispensing the medication will be aware of the study IDs in relation to the patient identity, in order to be able to dispense the test drug or the placebo per their assigned status as test or control subjects.

Study Drug and Placebo. Processed SFN-rich extract will be purchased in form of caplets from Nutramax Laboratories, Inc. 2208 Lakeside Blvd Edgewood, MD 21040. Caplets containing SFN-rich broccoli sprout extracts or microcrystalline cellulose (placebo) also from Nutramax Labs will be dispensed to participants in sealed bottles with instructions to keep them in a household freezer. Size of the caplet will be about the size of a 1000 mg Vit C pill (about 2 cm in length). The participants will be dosed, based on weight, in a double-blind fashion with identical appearing placebo or SFN caplets in a daily dose for 12 weeks of: two caplets for individuals <100 lb., three caplets for individuals 100-200 lb. and four caplets for individuals >200 lb. Avmacol Extra Strength or placebo will be prescribed by Dr. Jones and Philipovskiy and will be dispensed by local pharmacy or study coordinators at TTUHSC/UMC Lubbock. The investigators will be doing pill counts to make sure that volunteers have used as directed. The investigators will measure the Sulforaphane level in plasma by well-established method. 26 The drug and the placebo will be stored at the South West Cancer Center pharmacy based on manufacturer based guidelines and dispensed to each participant at their baseline visit then at DOX infusion visits 1, 2, and 3. Patients will be expected to maintain at least an 80% adherence to the medication regimen, in the absence of prohibitive toxicity. Adherence will be monitored through therapeutic drug level (Plasma sulforaphane levels of 120 ng/ml) monitoring as mentioned above and pill counts. For subjects who do not meet 80% compliance, they will be instructed on the importance of taking the pills as directed, but if their next visit demonstrates less than 80% compliance, they will be withdrawn from the study. As long as participants complete their 4th cycle of DOX chemotherapy treatment the investigators will still use their study data during analysis. If side effects are noted, patient will be asked to notify the study team of the same and will be evaluated within a suitable time frame based on severity of side effects.

SFN is a safe natural isolate. Above doses (30mg/caplet) are considered adequate to maintain intended therapeutic drug levels, while maintaining a simple study design and without significant concerns for drug toxicity It has been used in several clinical trials from doses ranging from 2-200 µmol/day for 2-28 weeks in 25-80 years old subjects without significant side-effects or toxicity (https://clinicaltrials.gov/ct2/results?term=sulforaphane&Search=Search), yet never in combination with DOX.

Statistical Considerations Data for the primary endpoint (DOX cardiotoxicity) and other binary outcomes will be summarized by treatment arm as number and proportion per arm. The change in DOX-cardiotoxicity rate with SFN compared to placebo will be assessed with a 1-sided Z-test (see Sample-size justification). Tumor size, plasma cardiac biomarkers, cardiac ejection fraction, DOX metabolite levels will be summarized by treatment arm and time point as means and standard deviations and graphed as box plots and profile plots. The investigators will adhere to ANOVA distributional assumptions so that appropriate data transformations can be applied. Data for each continuous variable will be analyzed for differences in group means at each time point with ANOVA or Mann-Whitney-Wilcoxon non-parametric tests at each time point. These tests will employ a more-stringent alpha = 0.02 significance level to adjust for the multiple comparisons without overinflating type II error. For subjects withdrawn from the study or do not complete the study for any reason, as long as they completed their 4th cycle of DOX chemotherapy treatment the investigators will still use their study data during analysis.

Sample-size justification. The number of subjects (35 per treatment arm; 70 total; the investigators expect some attrition, which this sample size addresses) is based on the primary endpoint of DOX-induced cardiac dysfunction, the rate of which was recently observed at our previous institution (UAMS) to be ~25%1. The investigators expect that SFN will decrease this to 5%. The cardiotoxicity rates for each arm will be compared via 1-sided pooled-variance Z-test at an alpha = 0.10. The statistical power of this test, conducted as described, needs to exceed 80% in order for our study to be generally recognized as having adequate statistical power. Our sample size provides the 1-sided pooled-variance Z-test with 83.2% power at 10% alpha to detect the expected 20-point decrease in DOX-toxicity rates from 25% in the placebo arm to 5% in the SFN arm.

The formal consent of each subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 89 years
2. No prior diagnosis of coronary artery, carotid artery or peripheral artery disease
3. Not pregnant or breastfeeding (urine pregnancy test will be done if female of childbearing potential)
4. Breast cancer requiring treatment with DOX-containing regimen above
5. Women in child bearing age group (18-50 years) will agree to use birth control for duration of study
6. Study subjects must be willing and able to swallow caplets, up to 8 daily.

Exclusion Criteria:

1. Currently on a research study with an investigational drug, or has been on one in the previous 30 days
2. Pregnant (by urine pregnancy test)
3. Baseline ejection fraction of less than 50%, evidence of left ventricular hypertrophy or baseline EKG reported as abnormal per cardiologist.
4. Inability to provide informed consent.
5. Prior history of chest radiation therapy
6. Diabetes or Hypertension or prior Myocardial infarction
7. Trastuzumab patients
8. Routinely taking vegetable or fruit-containing supplement pills (antioxidant phytochemicals) (daily vitamin pills ok)
9. Inability to follow up for safety monitoring
10. Prisoners
11. Previous or current use of cocaine or any illicit drug
12. Unable or unwilling to provide blood samples
13. Taking medications known to have cardiac effects, such as but not limited to, beta blockers, anti-arrhythmic agents, non dihydropyridine calcium channel blockers, ace inhibitors, NSAIDS, diuretic agents.
14. Unable to follow the protocol
15. Inability to receive anthracycline due to any reason (underlying baseline cardiac dysfunction due to other reasons, with an EF under 50%)
16. Patients already taking SFN OTC

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac function after DOX therapy with or without sulforaphane through diagnostic studies | At baseline and 1 year from baseline assessment.
  2D Echo will be used to measure cardiac function amongst patients on DOX therapy who are exposed to sulforaphane or placebo.

SECONDARY OUTCOMES:
Elevation of troponin levels as a surrogate evidence of DOX related cardiotoxicity will be checked at baseline, prior to each DOX therapy and then at 1 year from baseline assessment (Each cycle is 14 days). | At baseline, prior to each cycle of DOX, at completion of 4th cycle of DOX therapy and 1 year from baseline assessment.
  Troponin will be used to assess for cardiotoxicity amongst patients on DOX therapy who are exposed to sulforaphane or placebo.
Tumor size in patients on DOX therapy with or without sulforaphane treatment will be assessed at baseline, at completion of DOX chemotherapy (4 cycles planned with each cycle being 14 days) and at 1 year from baseline assessment. | 2 days before first DOX treatment, 2 days after completion of 4th cycle of DOX therapy and 1 year from first DOX treatment
  We will use PET imaging for comparison of change in tumor size for patients on DOX therapy with or without sulforaphane.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data generated from this project will be disseminated across the scientific community as rapidly as possible while adhering to the NIH Grants Policy on Availability of Research Results: Publications, Intellectual Property Rights, and Sharing Research Resources, issued in November 2016. The data will be available in password protected files, accessible only to investigators and with read only access to the databases. We will follow the guidelines established by NIH for Data Sharing Policy and Implementation and will ensure that all NIH privacy protection procedures are followed. We will make the dataset available to qualified investigators within 6 months of acceptance of the manuscript describing the main study findings. Investigators who request to use the dataset will be required to obtain IRB approval and to sign a data use agreement form before release of the data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: one year after completion of the study
Access Criteria: data will be provided upon request

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT03934905/Prot_SAP_001.pdf
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT03934905/ICF_000.pdf